CLINICAL TRIAL: NCT02464787
Title: Evaluation of Changes in Skin Carotenoid Score in Medical Students Following a Dietary Supplement-based Intervention
Brief Title: Evaluation of Changes in Skin Carotenoid Scores in Medical Students Following a Dietary Supplement-based Intervention
Acronym: SCS2015
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: L15-148; CRI 15-054 (Other: TTUHSC Clinical Research Institute)
Record Dates: First submitted 2015-05-28; First posted 2015-06-08 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Health Behavior
Keywords: antioxidants; carotenoids; diet
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Medical Students (Experimental): Medical students willing to maintain the increased consumption of LifePak Nano dietary supplements, two twin-sachet packets of seven (7) supplements twice per day, for the entire eight-week experimental period, to maintain the logs and to report at each of the times that measurements will be made.
  Interventions: Dietary Supplement: LifePak Nano

INTERVENTIONS:
Dietary Supplement: LifePak Nano — Two twin-sachet packets of seven (7) supplements twice per day, for the entire eight-week experimental period.

SUMMARY:
Skin Carotenoid Scores (SCS) are a biomarker of overall antioxidant status. This study extends an earlier study in which an increase in skin carotenoid scores (SCS) was observed in subjects who increased their intake of fruits and vegetables. The scores were determined using the Raman Spectroscopy. In that study subjects were assigned to one of four groups based on their baseline SCS. For unknown reasons, the groups with the highest and lowest baseline SCS failed to show an increase whereas the two intermediate groups did. One possible explanation might be that intakes varied more than expected and was not obvious due to self-reporting of intake of fruits and vegetables with different contents.

DETAILED DESCRIPTION:
This current project will be an interventional, non-invasive study examining changes in skin carotenoid levels over time in individuals who increase their carotenoid intake by taking a dietary supplement containing a known amount of carotenoids. After a two-week control period eating their normal diet, forty medical students meeting study inclusion criteria will be asked to take a dietary supplement over an eight week period of time. Students will be given twin-sachet packets of LifePak Nano supplements containing five capsules (dry ingredients) and two CR-6 Liponutrient softgel capsules (liquid ingredients, including omega-3 fatty acids and nanosized carotenoids). These will be taken twice a day with eight ounces of liquid at the morning and evening meal. SCS will be measured every 2 weeks. At the end of this period, the students will be asked to discontinue dietary supplement intake and follow their usual diet for 2 weeks then their SCS measured again.

ELIGIBILITY:
Inclusion Criteria:

1. Medical students must be willing to maintain the increased consumption of dietary supplements, two twin-sachet packets of seven (7) supplements twice per day, for the entire eight-week experimental period, to maintain the logs and to report at each of the times that measurements will be made. Individuals taking non-Pharmanex dietary supplements e.g. vitamins, minerals, herbals, and/or antioxidants will be asked to discontinue use at the time of the consenting to the study. Study supplements will replace all previous dietary supplements.
2. BMI between 20 and 29.9
3. Non-smoker, non-pregnant, non-lactating
4. No use of tanning beds or sunless tanning products during the study

Exclusion Criteria:

1. Prior participation in the previous study (L14 -128)
2. Individuals suffering from any chronic illness requiring ongoing medication, such as diabetes, hypertension, heart disease, GI disorders or other metabolic disorders
3. Individuals allergic or intolerant to shellfish,
4. pregnant or lactating women,
5. smokers
6. individuals with BMI > 30
7. Prior ingestion of LifePak Nano or other Pharmanex dietary supplements within the past 3 months.
8. SCS score less than 10,000 (< 10,000)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-03-20 (Actual); Study Completion 2016-10-14 (Actual)

PRIMARY OUTCOMES:
Change in skin carotenoid scores (SCS) | 12 weeks
  Skin Carotenoid Scores (SCS) are a biomarker of overall antioxidant status. The purpose of this study is to measure changes in SCS in medical students taking dietary supplements over a 12-week period of time. SCS will measured using a Bio-photonic Scanner. This scanner non-invasively measures carotenoid levels in the skin using optical signals. By placing the palm of the hand in front of a low-energy blue light for less than two minutes, the scanner can determine the SCS.

SECONDARY OUTCOMES:
Change in body weight | 12 weeks
  Weight will be measured on a calibrated balance scale over a 12-week period of time. Subjects will remove shoes, keys, cellphones, or other objects from their person before being weighed.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine B Chauncey, PhD, RDN, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

REFERENCES:
- [Background] Baranowski T. Understanding the behavioral linkages needed for designing effective interventions to increase fruit and vegetable intake in diverse populations. J Am Diet Assoc. 2011 Oct;111(10):1472-5. doi: 10.1016/j.jada.2011.07.014. No abstract available. PMID 21963012
- [Background] Dietary Guidelines for Americans, 2010; United States Department of Agriculture (USDA), United States Department of Health and Human Services: Dietary Guidelines for Americans, 2010. www.dietaryguidelines.gov
- [Background] Ermakov IV, Ermakova MR, McClane RW, Gellermann W. Resonance Raman detection of carotenoid antioxidants in living human tissues. Opt Lett. 2001 Aug 1;26(15):1179-81. doi: 10.1364/ol.26.001179. PMID 18049555
- [Background] Ermakov IV, Sharifzadeh M, Ermakova M, Gellermann W. Resonance Raman detection of carotenoid antioxidants in living human tissue. J Biomed Opt. 2005 Nov-Dec;10(6):064028. doi: 10.1117/1.2139974. PMID 16409093
- [Background] Ermakov IV, Gellermann W. Validation model for Raman based skin carotenoid detection. Arch Biochem Biophys. 2010 Dec 1;504(1):40-9. doi: 10.1016/j.abb.2010.07.023. Epub 2010 Aug 1. PMID 20678465
- [Background] Institute of Medicine (US) Panel on Dietary Antioxidants and Related Compounds. Dietary Reference Intakes for Vitamin C, Vitamin E, Selenium, and Carotenoids. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK225483/ PMID 25077263
- [Background] Jahns L, Johnson LK, Mayne ST, Cartmel B, Picklo MJ Sr, Ermakov IV, Gellermann W, Whigham LD. Skin and plasma carotenoid response to a provided intervention diet high in vegetables and fruit: uptake and depletion kinetics. Am J Clin Nutr. 2014 Sep;100(3):930-7. doi: 10.3945/ajcn.114.086900. Epub 2014 Jul 9. PMID 25008856
- [Background] Krebs-Smith SM, Guenther PM, Subar AF, Kirkpatrick SI, Dodd KW. Americans do not meet federal dietary recommendations. J Nutr. 2010 Oct;140(10):1832-8. doi: 10.3945/jn.110.124826. Epub 2010 Aug 11. PMID 20702750
- [Background] Mayne ST, Cartmel B, Scarmo S, Lin H, Leffell DJ, Welch E, Ermakov I, Bhosale P, Bernstein PS, Gellermann W. Noninvasive assessment of dermal carotenoids as a biomarker of fruit and vegetable intake. Am J Clin Nutr. 2010 Oct;92(4):794-800. doi: 10.3945/ajcn.2010.29707. Epub 2010 Aug 4. PMID 20685953
- [Background] Mayne ST, Cartmel B, Scarmo S, Jahns L, Ermakov IV, Gellermann W. Resonance Raman spectroscopic evaluation of skin carotenoids as a biomarker of carotenoid status for human studies. Arch Biochem Biophys. 2013 Nov 15;539(2):163-70. doi: 10.1016/j.abb.2013.06.007. Epub 2013 Jun 30. PMID 23823930
- [Background] McKay DL, Perrone G, Rasmussen H, Dallal G, Hartman W, Cao G, Prior RL, Roubenoff R, Blumberg JB. The effects of a multivitamin/mineral supplement on micronutrient status, antioxidant capacity and cytokine production in healthy older adults consuming a fortified diet. J Am Coll Nutr. 2000 Oct;19(5):613-21. doi: 10.1080/07315724.2000.10718959. PMID 11022875
- [Background] Scarmo S, Cartmel B, Lin H, Leffell DJ, Ermakov IV, Gellermann W, Bernstein PS, Mayne ST. Single v. multiple measures of skin carotenoids by resonance Raman spectroscopy as a biomarker of usual carotenoid status. Br J Nutr. 2013 Sep 14;110(5):911-7. doi: 10.1017/S000711451200582X. Epub 2013 Jan 28. PMID 23351238